CLINICAL TRIAL: NCT00514488
Title: A Phase III Study Comparing Imatinib Standard Dose (400 mg/Day) Versus Imatinib High Dose (800 mg/Day) in the Treatment of Newly Diagnosed High Risk Chronic Myeloid Leukemia in Chronic Phase
Brief Title: Imatinib Standard Dose (400 mg/Day) Versus Imatinib High Dose (800 mg/Day)
Acronym: CML022
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bologna (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ICSG/CML022
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2007-08-10 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Myeloid Leukemia
Keywords: chronic myeloid leukemia; STI 571; CML022
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: STI571 (400 mg/day; or 800 mg/day)

SUMMARY:
This is a phase III multicenter, open-label study designed to investigate the efficacy (hematological response, cytogenetic response and molecular response) and feasibility (tolerance, compliance and safety) of the tyrosine kinase inhibitor imatinib mesylate (formerly STI 571, GLIVEC, Novartis Pharma) at conventional dose (400 mg/daily) if compared with high dose (800 mg/daily) (serial number protocol ICSG/CML/022) in patients with Ph+ chronic myeloid leukemia (CML) in chronic phase (CP) previously untreated, at high Sokal risk.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=18 years
2. First chronic phase, less than 6 months of duration
3. High Sokal's risk
4. Ph positive
5. No previous treatment or hydroxiurea only.
6. Performance status (ECOG/WHO) < 2
7. Written informed consent

Exclusion Criteria:

1. Age <18
2. Low or intermediate Sokal risk score.
3. More than 6 months from diagnosis.
4. Second chronic, accelerated or blastic phase
5. Scheduled allogeneic stem cell transplantation within 1 year from diagnosis.
6. Performance status (ECOG/WHO) > 2
7. Inability to provide written informed consent
8. Pregnancy
9. Formal refusal of any recommendation of a safe contraception
10. Alcohol or drug addiction
11. Altered hepatic or renal function as defined by AST/ALT or bilirubine > 3 times upper normal limits (UNL) and by creatinine > 20mg/L
12. Any other disease or condition that by the advise of the responsible physician would make the treatment dangerous for the patient or would make the patient ineligible for the study, including physical, psychiatric, social and behavioural problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-06

PRIMARY OUTCOMES:
To determine the rate of complete cytogenetic response at 12 months in adult patients with previously untreated high Sokal risk CML treated with imatinib at 2 different dose levels of 400 and 800 mg/daily.

SECONDARY OUTCOMES:
The rate of major cytogenetic response,the kinetic and duration of cytogenetic response, the time to accelerated and blast crisis and overall survival,safety and tolerability of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, MD, Principal Investigator — Istituto di Ematologia e Oncologia Medica "L. e A. Seràgnoli" Università degli Studi di Bologna
Locations (1):
- Istituto di Ematologia e Oncologia Medica "L. e A. Seràgnoli", Bologna, Italy

REFERENCES:
- [Derived] Gugliotta G, Castagnetti F, Breccia M, Albano F, Iurlo A, Intermesoli T, Abruzzese E, Levato L, D'Adda M, Pregno P, Cavazzini F, Stagno F, Martino B, La Barba G, Sora F, Tiribelli M, Bigazzi C, Binotto G, Bonifacio M, Caracciolo C, Soverini S, Foa R, Cavo M, Martinelli G, Pane F, Saglio G, Baccarani M, Rosti G; Gruppo Italiano Malattie Ematologiche dell'Adulto - Chronic Myeloid Leukemia Working Party. Incidence of second primary malignancies and related mortality in patients with imatinib-treated chronic myeloid leukemia. Haematologica. 2017 Sep;102(9):1530-1536. doi: 10.3324/haematol.2017.169532. Epub 2017 Jun 1. PMID 28572163
- [Derived] Castagnetti F, Gugliotta G, Baccarani M, Breccia M, Specchia G, Levato L, Abruzzese E, Rossi G, Iurlo A, Martino B, Pregno P, Stagno F, Cuneo A, Bonifacio M, Gobbi M, Russo D, Gozzini A, Tiribelli M, de Vivo A, Alimena G, Cavo M, Martinelli G, Pane F, Saglio G, Rosti G; GIMEMA CML Working Party. Differences among young adults, adults and elderly chronic myeloid leukemia patients. Ann Oncol. 2015 Jan;26(1):185-192. doi: 10.1093/annonc/mdu490. Epub 2014 Oct 30. PMID 25361995
- [Derived] Luatti S, Castagnetti F, Marzocchi G, Baldazzi C, Gugliotta G, Iacobucci I, Specchia G, Zanatta L, Rege-Cambrin G, Mancini M, Abruzzese E, Zaccaria A, Grimoldi MG, Gozzetti A, Ameli G, Capucci MA, Palka G, Bernasconi P, Palandri F, Pane F, Saglio G, Martinelli G, Rosti G, Baccarani M, Testoni N; Gruppo Italiano Malattie Ematologiche dell'Adulto (GIMEMA) Working Party on CML. Additional chromosomal abnormalities in Philadelphia-positive clone: adverse prognostic influence on frontline imatinib therapy: a GIMEMA Working Party on CML analysis. Blood. 2012 Jul 26;120(4):761-7. doi: 10.1182/blood-2011-10-384651. Epub 2012 Jun 12. PMID 22692507
- [Derived] Gugliotta G, Castagnetti F, Palandri F, Breccia M, Intermesoli T, Capucci A, Martino B, Pregno P, Rupoli S, Ferrero D, Gherlinzoni F, Montefusco E, Bocchia M, Tiribelli M, Pierri I, Grifoni F, Marzocchi G, Amabile M, Testoni N, Martinelli G, Alimena G, Pane F, Saglio G, Baccarani M, Rosti G; Gruppo Italiano Malattie Ematologiche dell'Adulto CML Working Party. Frontline imatinib treatment of chronic myeloid leukemia: no impact of age on outcome, a survey by the GIMEMA CML Working Party. Blood. 2011 May 26;117(21):5591-9. doi: 10.1182/blood-2010-12-324228. Epub 2011 Mar 30. PMID 21450900
- [Derived] Marzocchi G, Castagnetti F, Luatti S, Baldazzi C, Stacchini M, Gugliotta G, Amabile M, Specchia G, Sessarego M, Giussani U, Valori L, Discepoli G, Montaldi A, Santoro A, Bonaldi L, Giudici G, Cianciulli AM, Giacobbi F, Palandri F, Pane F, Saglio G, Martinelli G, Baccarani M, Rosti G, Testoni N; Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Working Party on Chronic Myeloid Leukemia. Variant Philadelphia translocations: molecular-cytogenetic characterization and prognostic influence on frontline imatinib therapy, a GIMEMA Working Party on CML analysis. Blood. 2011 Jun 23;117(25):6793-800. doi: 10.1182/blood-2011-01-328294. Epub 2011 Mar 29. PMID 21447834
- [Derived] Testoni N, Marzocchi G, Luatti S, Amabile M, Baldazzi C, Stacchini M, Nanni M, Rege-Cambrin G, Giugliano E, Giussani U, Abruzzese E, Kerim S, Grimoldi MG, Gozzetti A, Crescenzi B, Carcassi C, Bernasconi P, Cuneo A, Albano F, Fugazza G, Zaccaria A, Martinelli G, Pane F, Rosti G, Baccarani M. Chronic myeloid leukemia: a prospective comparison of interphase fluorescence in situ hybridization and chromosome banding analysis for the definition of complete cytogenetic response: a study of the GIMEMA CML WP. Blood. 2009 Dec 3;114(24):4939-43. doi: 10.1182/blood-2009-07-229864. Epub 2009 Oct 1. PMID 19797518
- [Derived] Baccarani M, Rosti G, Castagnetti F, Haznedaroglu I, Porkka K, Abruzzese E, Alimena G, Ehrencrona H, Hjorth-Hansen H, Kairisto V, Levato L, Martinelli G, Nagler A, Lanng Nielsen J, Ozbek U, Palandri F, Palmieri F, Pane F, Rege-Cambrin G, Russo D, Specchia G, Testoni N, Weiss-Bjerrum O, Saglio G, Simonsson B. Comparison of imatinib 400 mg and 800 mg daily in the front-line treatment of high-risk, Philadelphia-positive chronic myeloid leukemia: a European LeukemiaNet Study. Blood. 2009 May 7;113(19):4497-504. doi: 10.1182/blood-2008-12-191254. Epub 2009 Mar 4. PMID 19264678